CLINICAL TRIAL: NCT06458647
Title: The Effect of Video Streaming With Virtual Reality on Anxiety, Comfort and Patient Satisfaction Before Coronary Angiography
Brief Title: The Effect of Video Streaming With Virtual Reality Before Coronary Angiography
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Associate Prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/581
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Anxiety; Comfort; Patient Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Individuals in the intervention group will be shown a video with virtual reality glasses before entering the angiography procedure.
  Interventions: Other: Video Streaming with Virtual Reality
- Control group (No Intervention): No application will be made to the control group before the procedure.

INTERVENTIONS:
Other: Video Streaming with Virtual Reality — In the study, patients in the intervention group will be watched videos of natural landscapes such as mountains, beaches and waterfalls with virtual reality goggles before the angiography procedure.
  Arms: Intervention group

SUMMARY:
This study was planned as a randomized controlled experimental study to examine the effects of virtual reality video on anxiety, comfort and patient satisfaction before coronary angiography. Data will be collected using the Descriptive Characteristics Questionnaire, State-Trait Anxiety Inventory, Early Postoperative Comfort Scale, Visual Analog Scale (VAS) for patient satisfaction and pain, Vital Signs Follow-up Form and Complication Follow-up Form.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled experimental study to examine the effects of virtual reality video on anxiety, comfort and patient satisfaction before coronary angiography. Data will be collected using the Descriptive Characteristics Questionnaire, State-Trait Anxiety Inventory, Early Postoperative Comfort Scale, Visual Analog Scale (VAS) for patient satisfaction and pain, Vital Signs Follow-up Form and Complication Follow-up Form. In addition to the standard practices of the clinic, individuals in the intervention group will be shown a video with virtual reality glasses before entering the angiography procedure. Only standard practices of the clinic will be applied to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Can speak and understand Turkish,
* Over 18 years of age,
* No previous angiography procedure,
* Oriented to place and time,
* No psychiatric illness,
* Not taking any sedative medication,
* No vision and hearing problems,
* Patients who volunteered to participate in the study will be included.

Exclusion Criteria:

* Patients with any pain or chronic pain prior to coronary angiography,
* Patients diagnosed with anxiety,
* Patients with pacemakers,
* Patients requiring emergency angiography,
* Patients taking antihistamines and psychiatric drugs,
* Patients who did not volunteer to participate in the study,
* Patients taking tranquilizers or pain medication up to 5 hours before the angiography procedure were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 30 minutes after angiography
  This inventory, which consists of a total of 40 items, is analyzed in two separate sections: The first part is the State Anxiety Inventory, which consists of 20 items, and the individual answers this section with his/her current feelings. The second part is the Trait Anxiety Inventory, which also consists of 20 items, and the individual answers this section with the feelings they have felt in the last 7 days.
Comfort | 30 minutes after angiography
  The scale, which is based on the concept of comfort, consists of a total of 24 items, 12 of which question the comfort status of the individual before and after the surgical intervention, 12 of which question positive and 12 of which question negative experiences.
Patient satisfaction | 30 minutes after angiography
  Patients will be asked to rate their satisfaction with the intervention on a 10-point scale.

IPD SHARING:
Plan to Share IPD: No